CLINICAL TRIAL: NCT07315841
Title: A Prospective Study Evaluating the Accuracy of Indocyanine Green Fluorescence Imaging in Detecting Lesions During Tenosynovial Giant Cell Tumor Surgery
Brief Title: Accuracy of Indocyanine Green (ICG) Fluorescence Imaging in Tenosynovial Giant Cell Tumor Surgery
Acronym: ICG-TGCT
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Shanghai Jiao Tong University Affiliated Sixth People's Hospital (Other)
Responsible Party: Principal Investigator, Qingcheng Yang, Chief Orthopaedic Surgeon & Director, Shanghai Jiao Tong University Affiliated Sixth People's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2025-147; 2025-147 (Other: Ethics Committee of Shanghai Sixth People's Hospital)
Record Dates: First submitted 2025-12-19; First posted 2026-01-02 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2026-01

CONDITIONS: Tenosynovial Giant Cell Tumor
Keywords: Indocyanine Green; Fluorescence Imaging; Near-Infrared Imaging; Tenosynovial Giant Cell Tumor
MeSH Terms: conditions — Giant Cell Tumor of Tendon Sheath | interventions — Indocyanine Green

STUDY DESIGN:
Intervention Model Description: This is a prospective, single-center, single-arm study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ICG Fluorescence Imaging Group (Experimental): All enrolled participants receive ICG fluorescence-guided surgery. Following standard tumor resection, the surgical bed is systematically explored using a near-infrared fluorescence imaging system. The intervention consists of detecting residual fluorescence signals, obtaining verification samples for pathology, and performing supplementary resection of confirmed suspicious lesions to achieve potentially cleaner surgical margins.
  Interventions: Drug: Indocyanine Green

INTERVENTIONS:
Drug: Indocyanine Green — Participants receive an intravenous injection of Indocyanine Green (ICG) at a dose of 0.25-0.5 mg/kg, 1-3 hours prior to surgery. Intraoperatively, a near-infrared fluorescence imaging system is used to guide the exploration. The intervention involves a "verify first, treat later" protocol: it includes diagnostic verification sampling of fluorescence-positive areas and, crucially, therapeutic supplementary resection of residual fluorescent lesions that were missed during standard white-light surgery.

SUMMARY:
This study evaluates the diagnostic accuracy of Indocyanine Green (ICG) fluorescence imaging in visualizing Tenosynovial Giant Cell Tumor (TGCT) lesions during surgery. Patients diagnosed with TGCT will receive an intravenous injection of ICG prior to the operation to label tumor tissues. During the procedure, surgeons will use a near-infrared fluorescence imaging system to visualize the tumor and potential residual lesions in the surgical bed. The study aims to determine the sensitivity, specificity, positive predictive value, and negative predictive value of ICG fluorescence imaging by comparing the intraoperative fluorescence findings with the final pathological results of the resected tissues.

DETAILED DESCRIPTION:
Tenosynovial Giant Cell Tumor (TGCT), especially the diffuse type, poses a significant surgical challenge due to its infiltrative growth and high recurrence rate. This prospective, single-center, single-arm study aims to evaluate the accuracy of Indocyanine Green (ICG) fluorescence imaging in visualizing TGCT lesions during surgery. Eligible patients will receive an intravenous injection of ICG (0.25-0.5 mg/kg) 1-3 hours before surgery. Following standard tumor resection under white light, the surgical bed will be systematically explored using a near-infrared fluorescence imaging system to visualize potential tumor tissues. The surgeon will obtain validation samples from both fluorescence-positive areas and fluorescence-negative background tissues for blinded pathological assessment. The study will quantify the diagnostic performance of ICG imaging by calculating sensitivity, specificity, positive predictive value, and negative predictive value based on the pathological gold standard, alongside secondary analyses of tumor-to-background ratios and microscopic tumor boundary concordance.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with Tenosynovial Giant Cell Tumor (TGCT), including both Localized-type (L-TGCT) and Diffuse-type (D-TGCT), via preoperative biopsy or typical imaging (MRI), and scheduled for surgical resection.
* Capable of understanding the study and voluntarily signing the written informed consent form.

Exclusion Criteria:

* Known severe history of allergy to Indocyanine Green (ICG) or iodine.
* Severe liver dysfunction.
* Women who are pregnant or lactating.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2026-01-02 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Diagnostic Accuracy of ICG Fluorescence Imaging (Sensitivity, Specificity, PPV, NPV) | From the time of surgery until the final pathology report is available, assessed up to 1 week post-operatively.
  The diagnostic performance of ICG fluorescence imaging in detecting TGCT lesions will be evaluated by comparing the intraoperative fluorescence status (Positive/Negative) with the final histopathological diagnosis (Tumor/Non-tumor) of the resected specimens. The unit of analysis is the individual specimen. The following metrics will be calculated: Sensitivity, Specificity, Positive Predictive Value (PPV), and Negative Predictive Value (NPV).

SECONDARY OUTCOMES:
Tumor-to-Background Ratio (TBR) | Intraoperative
  TBR is a quantitative measure of fluorescence intensity. It will be calculated by dividing the mean fluorescence intensity of the tumor region by the mean fluorescence intensity of the adjacent normal background tissue using image analysis software. Values will be compared between Diffuse-type TGCT (D-TGCT) and Localized-type TGCT (L-TGCT) cohorts.
Incidence of ICG-Related Adverse Events | From the time of ICG injection through 24 hours post-surgery
  The number of participants experiencing adverse events related to ICG administration (e.g., allergic reactions, anaphylactic shock) will be monitored and recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Sixth People's Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Nicoli F, Saleh DB, Baljer B, Chan CD, Beckingsale T, Ghosh KM, Ragbir M, Rankin KS. Intraoperative Near-infrared Fluorescence (NIR) Imaging With Indocyanine Green (ICG) Can Identify Bone and Soft Tissue Sarcomas Which May Provide Guidance for Oncological Resection. Ann Surg. 2021 Feb 1;273(2):e63-e68. doi: 10.1097/SLA.0000000000003857. PMID 32224746
- [Result] Wang H, Ji T, Qu H, Yan T, Li D, Yang R, Tang X, Guo W. Indocyanine green fluorescence imaging may detect tumour residuals during surgery for bone and soft-tissue tumours. Bone Joint J. 2023 May 1;105-B(5):551-558. doi: 10.1302/0301-620X.105B5.BJJ-2022-0803.R1. PMID 37121591
- [Result] Huang H, He S, Wei R, Zhu X, Deng Z, Wang Y, Guo L, Lei J, Cai L, Xie Y. Near-infrared (NIR) imaging with indocyanine green (ICG) may assist in intraoperative decision making and improving surgical margin in bone and soft tissue tumor surgery. J Surg Oncol. 2023 Sep;128(4):612-627. doi: 10.1002/jso.27306. Epub 2023 May 13. PMID 37178368
- [Result] He K, Zhou J, Yang F, Chi C, Li H, Mao Y, Hui B, Wang K, Tian J, Wang J. Near-infrared Intraoperative Imaging of Thoracic Sympathetic Nerves: From Preclinical Study to Clinical Trial. Theranostics. 2018 Jan 1;8(2):304-313. doi: 10.7150/thno.22369. eCollection 2018. PMID 29290809
- [Result] He K, Li P, Zhang Z, Liu J, Liu P, Gong S, Chi C, Liu P, Chen C, Tian J. Intraoperative near-infrared fluorescence imaging can identify pelvic nerves in patients with cervical cancer in real time during radical hysterectomy. Eur J Nucl Med Mol Imaging. 2022 Jul;49(8):2929-2937. doi: 10.1007/s00259-022-05686-z. Epub 2022 Mar 1. PMID 35230489
- [Result] Vinegoni C, Botnaru I, Aikawa E, Calfon MA, Iwamoto Y, Folco EJ, Ntziachristos V, Weissleder R, Libby P, Jaffer FA. Indocyanine green enables near-infrared fluorescence imaging of lipid-rich, inflamed atherosclerotic plaques. Sci Transl Med. 2011 May 25;3(84):84ra45. doi: 10.1126/scitranslmed.3001577. PMID 21613624
- [Result] Newton AD, Predina JD, Shin MH, Frenzel-Sulyok LG, Vollmer CM, Drebin JA, Singhal S, Lee MK 4th. Intraoperative Near-infrared Imaging Can Identify Neoplasms and Aid in Real-time Margin Assessment During Pancreatic Resection. Ann Surg. 2019 Jul;270(1):12-20. doi: 10.1097/SLA.0000000000003201. PMID 31188797
- [Result] Gouin F, Noailles T. Localized and diffuse forms of tenosynovial giant cell tumor (formerly giant cell tumor of the tendon sheath and pigmented villonodular synovitis). Orthop Traumatol Surg Res. 2017 Feb;103(1S):S91-S97. doi: 10.1016/j.otsr.2016.11.002. Epub 2017 Jan 2. PMID 28057477
- [Result] Stacchiotti S, Durr HR, Schaefer IM, Woertler K, Haas R, Trama A, Caraceni A, Bajpai J, Baldi GG, Bernthal N, Blay JY, Boye K, Broto JM, Chen WT, Dei Tos PA, Desai J, Emhofer S, Eriksson M, Gronchi A, Gelderblom H, Hardes J, Hartmann W, Healey J, Italiano A, Jones RL, Kawai A, Leithner A, Loong H, Mascard E, Morosi C, Otten N, Palmerini E, Patel SR, Reichardt P, Rubin B, Rutkowski P, Sangalli C, Schuster K, Seddon BM, Shkodra M, Staals EL, Tap W, van de Rijn M, van Langevelde K, Vanhoenacker FMM, Wagner A, Wiltink L, Stern S, Van de Sande VM, Bauer S. Best clinical management of tenosynovial giant cell tumour (TGCT): A consensus paper from the community of experts. Cancer Treat Rev. 2023 Jan;112:102491. doi: 10.1016/j.ctrv.2022.102491. Epub 2022 Dec 6. PMID 36502615
- [Result] Palmerini E, Staals EL. Treatment updates on tenosynovial giant cell tumor. Curr Opin Oncol. 2022 Jul 1;34(4):322-327. doi: 10.1097/CCO.0000000000000853. PMID 35837703